CLINICAL TRIAL: NCT04598620
Title: Non-invasive Prognostication of COVID-19 Patients by Use of Biomarkers in Exhaled Breath Condensate
Acronym: VTE-COVID-19
Status: Completed | Type: Observational
Sponsor: Inger Lise Gade (Other)
Collaborators: Aarhus University Hospital Skejby (Other)
Responsible Party: Sponsor-Investigator, Inger Lise Gade, MD, PhD, Registrar, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Other Study IDs: ILG-VTE-COVID-19-2020; N-20200069 (Other: Den Videnskabsetiske Komite for Region Nordjylland)
Record Dates: First submitted 2020-10-21; First posted 2020-10-22 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Covid19; Corona Virus Infection
Keywords: Exhaled breath condensate
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Exhaled breath condensate (EBC) Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of this study is to assess if analysis of exhaled breath condensate (EBC) can provide useful prognostic markers for admission to the intensive care unit (ICU) due to acute respiratory insufficiency among patients with Coronavirus disease 2019 (COVID-19). Additionally, to give a characterization of the lung damage caused by COVID-19 by analysis of daily blood samples.

The hypothesis is that the protein content of the EBC from COVID-19 patients who require admission to the ICU differs from the EBC from COVID-19 patients with uncomplicated hospitalization, potentially providing diagnostic markers of COVID-19 related pulmonary damage.

DETAILED DESCRIPTION:
Two EBC samples will be collected from each study participant; a baseline sample (at admission) and a sample at either hospital discharge or transfer to the ICU. In addition, blood samples will be collected in order to investigate the pathophysiology of COVID-19 using metabolomics analysis, and for standardization and validation of the putative markers from the EBC.

The investigators will collect EBC from COVID-19 positive patients acutely admitted to Aalborg University Hospital due to COVID-19 symptoms and compare the protein and metabolite profiles in patients, who are treated at the ward with patients, who are transferred to the ICU for mechanical ventilation. The main-outcome (i.e. means of the relative amounts of specific proteins in the EBC samples) will be compared by unpaired t-tests after assessment of normality and standard deviations within the two groups in the following comparison: EBC collected at admission (baseline) from patients who did not need mechanical ventilation vs. EBC at admission from patients who did need mechanical ventilation. Paired t-tests will compare the proteins in baseline EBC samples and samples at either transfer to the ICU intubation or discharge to home in order to describe the pathophysiology in the two groups (no ICU need versus need of ICU admission). The investigators will not collect EBC from patients admitted to the ICU for open-circuit respiratory support, e.g. high-flow oxygenation; these patients will be asked to give an EBC sample before discharge, like the patients who did not need ICU care.

A blood sample will be drawn at the two days of EBC collection (i.e. a 9 mL tube drawn along with routine work-up blood samples) from the study participants for two purposes: 1) Standardization of the putative markers and verification and supplementing analysis of the EBC markers. In order to qualify the most suitable markers and substrates for standardization, the analysis of the EBC samples must be completed before the blood samples can be analyzed. Conventional biochemical analysis will be used for this purpose. 2) Pathophysiological description of patients hospitalized with COVID-19 using metabolomics and proteomics analysis. No genetic analysis will be conducted on the stored blood samples.

After collection of the EBC, the samples will be stored directly in the collection tube marked with study subject id at -80⁰C. The EBC samples will be used solely for the subsequent analysis of the protein composition (i.e. proteomics) and metabolites (i.e. metabolomics).

The collection of EBC will not lead to deviations from standard diagnostic procedures or treatments. The patients will have routine blood samples drawn as a part of the diagnostic work-up and daily disease monitoring. The investigators will ask for consent to draw an extra 9 mL blood sample along with the routine blood samples at the two days of EBC collection.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and admitted at Aalborg Hospital with confirmed COVID-19
* Need for hospitalization due to COVID-19 symptoms.
* Able to provide informed consent

Exclusion Criteria:

• Need for vasopressor therapy, mechanical ventilation, extracorporal circulation, or dialysis at admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 positive patients acutely admitted to Aalborg University Hospital due to COVID-19 symptoms.
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2020-09-19 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Prediction of admission to ICU in hospitalized COVID-19 patients | 1 year
  The primary outcome is prediction of admission to ICU in hospitalized COVID-19 patients by use of one or more novel biomarkers in the EBC

SECONDARY OUTCOMES:
Pathophysiology in COVID-19 patients | 1 year
  In a sub-study, we will collect the daily blood samples for analysis in order to investigate the pathophysiology in COVID-19, and for standardization and validation of putative EBC markers in the blood.

CONTACTS AND LOCATIONS:
Overall Officials: Inger L Gade, MD, PhD, Principal Investigator — Aalborg University Hospital
Locations (1):
- Aalborg Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gade IL, Bodilsen J, Mariager T, Hertz S, Duerlund LS, Holm CK, Madsen PH, Bennike TB, Honore B. Exhaled breath protein composition in patients hospitalised during the first wave of COVID-19. J Breath Res. 2025 May 16;19(3). doi: 10.1088/1752-7163/add617. PMID 40341493